CLINICAL TRIAL: NCT04164355
Title: Evaluation of Retinal and Choriocapillary Vascular Changes Using Optical Coherence Tomography Angiography in Patients Undergoing Tadalafil 20mg on Alternative Days: a Single-centre Prospective-control
Brief Title: Study of Retinal and Choriocapillary Vascular Changes in Patients Undergoing Tadalafil 20mg
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, Principal Investigator, Federico II University
Other Study IDs: PT1515/19
Record Dates: First submitted 2019-11-11; First posted 2019-11-15 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Erectile Dysfunction Following Radical Prostatectomy
MeSH Terms: interventions — Tadalafil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients undergoing Tadalafil: Patients after radical prostatectomy, undergoing Tadalafil 20 mg orally, on alternative days, for 6 months
  Interventions: Drug: Tadalafil 20 MG
- Control Group: Healthy controls without previous surgery of radical prostatectomy.

INTERVENTIONS:
Drug: Tadalafil 20 MG — To study retinal and choriocapillary features in patients undergoing Tadalafil 20 mg orally, on alternate days, at baseline and 1, 3, 6 months after radical prostatectomy
  Other Names: Cialis
  Groups: Patients undergoing Tadalafil

SUMMARY:
This study evaluates the retinal and choriocapillary vascular features in patients under the effects of Tadalafil 20mg using optical coherence tomography angiography.

DETAILED DESCRIPTION:
Tadalafil is a an inhibitor of the enzyme phosphodiesterase and it works by increasing blood flow to the penis thus promoting the erection.

This drug represents an treatment for erectile dysfunction in patients after radical prostatectomy.

The optical coherence tomography angiography represents a novel and non-invasive diagnostic technique that allows a detailed and quantitative analysis of retinal and choriocapillary vascular features.

The study evaluates the changes in optical coherence tomography angiography parameters at baseline and after 1, 3, 6 months after the somministration of Tadalafil 20 mg orally.

ELIGIBILITY:
Inclusion Criteria:

* age older than 45 years
* diagnosis of erectile dysfunction due to surgery of radical prostatectomy
* treatment-naïve with Tadalafil for erectile dysfunction
* absence of vitreoretinal and vascular retinal diseases
* absence of diabetes

Exclusion Criteria:

* age younger than 45 years
* diagnosis of erectile dysfunction due to other causes
* previous treatments before Tadalafil for erectile dysfunction
* presence of vitreoretinal and vascular retinal diseases
* presence of diabetes.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participans were older than 45 years with diagnosis of erectile dysfunction due to surgery of radical prostatectomy. They did not receive previous treatment before Tadalafil and they have not other ophthalmological disease and diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-07-04 (Actual); Primary Completion 2021-04-25 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
The measurements of retinal and choriocapillary vessel density in patients undergoing Tadalafil after radical prostatectomy | Six months
  Changes in retinal and choriocapilary vessel density in 40 patients undergoing Tadalafil 20 mg orally, on alternate days, at baseline and 1, 3, 6 months after radical prostatectomy, using optical coherence tomography angiography. The parameters analyzed by optical coherence tomography angiography were: retinal and choriocapillary vessel density

CONTACTS AND LOCATIONS:
Overall Officials: Gilda Cennamo, Principal Investigator — Federico II University
Locations (1):
- University of Naples "Federico II", Naples, Italy